CLINICAL TRIAL: NCT06066281
Title: Validation and Standardization of the Consecutive-Letter Substitution Task (CST) Test in an Italian Population Sample
Brief Title: Validation of the Consecutive-Letter Substitution Task (CST)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Prof. Massimo Filippi, Head of Neurology, IRCCS San Raffaele
Other Study IDs: VAL-CST
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers
Keywords: Processing Speed; Neuropsychological Tests; Reference Standards
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteers: 480 healthy subjects between the ages of 18 and 75, Italian native speakers, willing and able to comply with study procedures.
  Interventions: Behavioral: Neuropsychological assessment

INTERVENTIONS:
Behavioral: Neuropsychological assessment — All participants who will meet the inclusion criteria will be adminstered a pencil-paper neuropsychological tests battery including: the Digit Span Backward Task, the Brief Repeatable Battery of Neuropsychological Tests and the CST. After 15 days from the baseline evaluation the CST will be re-administrated to all subjects.

SUMMARY:
The CST is a new neuropsychological test created to measure information processing speed, which is frequently impaired in patients with multiple sclerosis. The aim of the study is to validate the CST through the administration on a representative sample of healthy subjects of the Italian population. Each subject will be administered a standardized battery of neuropsychological tests (Digit Span Task and Brief Repeatable Battery of Neuropsychological Tests which includes Selective Reminding Test, Spatial Recall Test, Symbol Digit Modalities Test, Paced Auditory Serial Addition Test and Word List Generation), and the CST in order to verify its validity. After 15 days from the baseline, the CST will be re-administrated to all subjects to assess the reliability of the test.

DETAILED DESCRIPTION:
STUDY DESIGN: This is a monocentric, observational study with low-risk intervention.

STUDY PROCEDURES: The CST consists of a standard A4 sheet of paper that shows 135 items within a table of nine rows by fifteen columns. The subject is timed to determine how many correct responses can be made in 90 seconds. The first ten items are administered without a time limit for familiarizing examinee with the task before proceeding with the actual test. The study will involve two evaluations:

1. Baseline, in which CST, the Digit Span Backward Task and the Brief Repeatable Battery of Neuropsychological Tests ([BRB-N] including Selective Reminding Test [SRT], Spatial Recall Test [SPART], Symbol Digit Modalities Test [SDMT], Paced Auditory Serial Addition Test [PASAT] and Word List Generation [WLG]) will be administered in order to perform a comparison between these tools useful for the validation analysis. Moreover, the Montgomery-Åsberg Depression Rating Scale (MADRS) will be administered to detect the presence of depressive symptoms which could affect cognitive performance;
2. Follow-up, after 15 days from the baseline, in which CST will be re-administrated to all subjects to assess the reliability of the test.

At baseline, all participants will be informed of the project purpose and will be asked whether they agree to participate signing the consent form, then the tests will be administered. The first evaluation will require approximately 45 minutes, whereas the second one will take around 5 minutes. The CST, BRB-N, Digit Span Backward Task and MADRS will be administered by trained psychologists.

COLLECTED VARABLES:

Demographic variables

- Age, sex and education.

Neuropsychological and psychological variables

In accordance with the objectives of the study, the neuropsychological and psychological variables collected will be:

* Verbal learning and delayed recall assessed with the SRT, included in the BRB-N. The SRT includes a list of 12 words and uses six consecutive learning trials and a delayed trial. A word recalled on two consecutive trials is considered to have entered long-term storage (LTS) on the first of these trials and scored as LTS on all following trials. The total sum of the words in LTS of all six trials is taken (SRT-LTS). If a word in LTS is consistently recalled on all subsequent trials, it is then scored as in Consistent Long Term Retrieval (CLTR). The total sum of the words in CLTR of all six trials is taken (SRT-CLTR). The Delayed Recall (SRT-D) is the total number of words recalled after the delayed period.
* Visuospatial learning and delayed recall assessed with the SPART, included in the BRB-N. In the test, a checkerboard, with ten checkers arranged in a particular pattern, is shown to the subject for ten seconds. Then, the subject is asked to reproduce the same pattern with ten checkers on an empty checkerboard. The test includes three consecutive trials and a delayed trial. The score is the total number of correct responses for the three trials (SPART) and the delayed recall trial (SPART-D).
* Attention and processing speed measured with the SDMT, included in the BRB-N.
* Sustained attention and speed of information processing assessed with PASAT, included in the BRB-N. The subject hears a series of single digit numbers from a cassette tape recorder that are presented at the rate of one every 3 seconds in the first part of the test (PASAT 3), or at the rate of one every 2 seconds in the second part (PASAT 2). The subject is asked to add each consecutive digit to the one immediately preceding it. Sixty-one digits are presented for each part and each part has a maximum of 60 correct answers. In the administration of this test, it should be considered that tapes tend to become slower over time: therefore, the use of compact-discs and compact-disc players should be favoured.
* Verbal fluency on semantic stimulus assessed with WLG, included in the BRB-N. The subject is asked to produce as many words as possible belonging to a semantic category (vegetables and fruits in version) within 90 seconds. The score is the number of correct words.
* Working memory assessed with Digit Span backward Task. The examiner pronounces a list of digits at a rate of approximately one digit per second and subjects are required to the sequence of digits in the reverse order. If they succeed, a list one digit longer is presented. If they fail, a second list of the same length is presented. If subjects are successful on the second list, a list one digit longer is given, as before. However, if subjects also fail on the second list, the test is ended. The length of the digit sequences gradually increases, starting with a sequence of two numbers to a sequence of maximum eight items. The span is established as the length of the longest list recalled correctly.
* Depressive symptoms assessed with MADRS. It is a 10-item depression scale. The items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts) were empirically selected to represent core symptoms of depressive disorders. There are seven levels for the scoring items, from 0 to 6. The final score is the sum of all items' scores. A score > 9 indicates the presence of clinically significant symptoms of depression.
* Information processing speed assessed with CST. The tool has been described above.

SAMPLE SIZE CALCULATION: The minimum sample size, needed to assure good recovery of population factors is not constant, but rather is dependent on some aspects of the variables and design in a given study. A sample size of at least 300 is required in case of low communalities and a small number of factors, while, the sample size needed for reliability studies is of a minimum of 400 subjects. On the other hand, taking into account a potential screen failure rate approximately 6% to 7% of the entire sample and a potential drop-out rate estimating it about 10% of the entire sample, 80 subjects were addedd in order to obtain a total sample size of approximately 480 healthy subjects. Finally, the 480-sample size planned in this project, based on indications from the literature, must be considered wide enough to respect statistical standard and follow the study purpose.

STUDY POPULATION: The objective is to recruit 480 healthy subjects, in order to have a sample wide enough to represent the Italian population. Some healthy subjects will be asked their willingness to participate to the study by general practitioners that are accredited with "San Raffaele Scientific Institute"; a cover letter explaining the project's purpose and the informed consent will be provided. Other subjects will be recruited directly from the healthy control population available to participate at research protocols of our Research Unit. Staff and students from the Vita-Salute San Raffaele University will also be recruited.

STATISTICAL CONSIDERATIONS: The first part of analysis will be focused on the validation of the CST, including reliability and validity processes, and principal component analysis. Convergent and discriminant construct validity will be estimated using a bivariate correlation between CST and the SRT, SPART, SDMT, PASAT, WLG and Digit Span Backward Task. In the second part of the analysis, a predictive analysis will be carried out to identify possible predictors of information processing speed level in healthy adults.

SAFETY: Neuropsychological evaluations at baseline and at follow-up will be performed as a standard of care and do not carry any risk since as they consist of paper-and-pencil tests.

ETHICAL AND REGULATORY CONSIDERATIONS: The study will be conducted in accordance with Good Clinical Practice (GCP), as defined by the International Conference on Harmonization (ICH), the World Health Organization (WHO), and any local directives and in compliance with the protocol. The protocol, any amendments, and the subject informed consent will receive Institutional Review Board/Independent Ethics Committee (IRB/IEC) approval/favorable opinion before initiation of the study. The personnel involved in the study will include people qualified by education, training, and experience to perform their respective tasks and the study will not use the services of study personnel for whom sanctions have been invoked or where there has been scientific misconduct or fraud. The Investigator(s) undertake(s) the responsibility to perform the study in accordance with this Protocol, GCP, and the applicable regulatory requirements. The Investigator is required to ensure compliance with the visit schedule and procedures required by the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Italian native speaker;
* No neurological and/or psychiatric diseases;
* Willing and able to comply with study procedures.

Exclusion Criteria:

* History of drug, alcohol or substance abuse;
* A score > 9 on the Montgomery-Åsberg Depression Rating Scale (MADRS), which is the lower limit for mild depressive symptoms;
* Any person unable to understand and follow the instructions of the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Four hundred and eighty healthy subjects will be recruited, in order to have a sample wide enough to represent the Italian population
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Test-retest reliability | 15 days
  CST intra-class correlation coefficients will be calculated on total CST scores which are expected to remain stable
Construct validity | 2 years
  CST covergent and discriminant construct validity: neuropsychological tests scores comparisons will be performed to investigate the concurrent convergent validity of the CST. Pearson correlation coefficients will be calculated to explore the association between CST scores and Selective Reminding Test (SRT), Spatial Recall Test (SPART), Symbol Digit Modalities Test (SDMT), Paced Auditory Serial Addition Test (PASAT) and Word List Generation (WLG) and Digit Span Backward Task scores. Exploratory and confirmatory factor analysis will be performed to determine latent variables.
Italian normative data | 2 years
  Multivariable hierarchical linear models will be performed to identify possible predictors (among demographic variables) of information processing speed assessed with the CST in healthy adults. A p-value <0.05 will be considered as significant. When a significant relationship between test scores and the variables is found, the regression coefficients will be used to adjust raw data. After correcting for the relevant demographic factors, the fifth percentile of CST scores distribution will be calculated to determine the cut-off value.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Filippi, MD, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
The dataset including all the data obtained from this study will be available from the Principal Investigator upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The dataset including all the data obtained from this study will be available 6 months after the publication of the results.
Access Criteria: The dataset including all the data obtained from this study will be available from the Principal Investigator upon reasonable request.

REFERENCES:
- [Background] Costa SL, Genova HM, DeLuca J, Chiaravalloti ND. Information processing speed in multiple sclerosis: Past, present, and future. Mult Scler. 2017 May;23(6):772-789. doi: 10.1177/1352458516645869. Epub 2016 May 9. PMID 27207446
- [Background] Benedict RH, DeLuca J, Phillips G, LaRocca N, Hudson LD, Rudick R; Multiple Sclerosis Outcome Assessments Consortium. Validity of the Symbol Digit Modalities Test as a cognition performance outcome measure for multiple sclerosis. Mult Scler. 2017 Apr;23(5):721-733. doi: 10.1177/1352458517690821. Epub 2017 Feb 16. PMID 28206827
- [Background] Monaco M, Costa A, Caltagirone C, Carlesimo GA. Forward and backward span for verbal and visuo-spatial data: standardization and normative data from an Italian adult population. Neurol Sci. 2013 May;34(5):749-54. doi: 10.1007/s10072-012-1130-x. Epub 2012 Jun 12. PMID 22689311
- [Background] Amato MP, Portaccio E, Goretti B, Zipoli V, Ricchiuti L, De Caro MF, Patti F, Vecchio R, Sorbi S, Trojano M. The Rao's Brief Repeatable Battery and Stroop Test: normative values with age, education and gender corrections in an Italian population. Mult Scler. 2006 Dec;12(6):787-93. doi: 10.1177/1352458506070933. PMID 17263008
- [Background] Zimmerman M, Chelminski I, Posternak M. A review of studies of the Hamilton depression rating scale in healthy controls: implications for the definition of remission in treatment studies of depression. J Nerv Ment Dis. 2004 Sep;192(9):595-601. doi: 10.1097/01.nmd.0000138226.22761.39. PMID 15348975
- [Background] MacCallum RC, Widaman KF, Preacher KJ, Hong S. Sample Size in Factor Analysis: The Role of Model Error. Multivariate Behav Res. 2001 Oct 1;36(4):611-37. doi: 10.1207/S15327906MBR3604_06. PMID 26822184
- [Background] Charter RA. Sample size requirements for precise estimates of reliability, generalizability, and validity coefficients. J Clin Exp Neuropsychol. 1999 Aug;21(4):559-66. doi: 10.1076/jcen.21.4.559.889. PMID 10550813
- [Background] Gigantesco A, Ferrante G, Baldissera S, Masocco M; PASSI coordinating group. Depressive Symptoms and Behavior-Related Risk Factors, Italian Population-Based Surveillance System, 2013. Prev Chronic Dis. 2015 Oct 29;12:E183. doi: 10.5888/pcd12.150154. PMID 26513439
- [Background] Sakpal TV. Sample size estimation in clinical trial. Perspect Clin Res. 2010 Apr;1(2):67-9. PMID 21829786
- [Background] Galinowski A, Lehert P. Structural validity of MADRS during antidepressant treatment. Int Clin Psychopharmacol. 1995 Sep;10(3):157-61. doi: 10.1097/00004850-199510030-00004. PMID 8675968